CLINICAL TRIAL: NCT04945980
Title: Manipulation of Beef Fatty Acids to Tailor Ground Beef Products to Individual Consumer Needs
Brief Title: Ground Beef and Cardiovascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB2005-0435
Record Dates: First submitted 2021-06-25; First posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Lipoprotein Metabolism Disorder
Keywords: ground beef; lipoprotein cholesterol; cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: A 2-period, randomized cross-over design was used. Each participant completed two 5-wk diet interventions in a randomly assigned order with a 4-wk washout period between the test diet interventions.
Who Masked: Participant
Masking Description: Participants were blinded to treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-MUFA ground beef (Experimental): Participants consumed ground beef low in monounsaturated fatty acids.
  Interventions: Dietary Supplement: Ground beef
- High-MUFA ground beef (Experimental): Participants consumed ground beef high in monounsaturated fatty acids.
  Interventions: Dietary Supplement: Ground beef

INTERVENTIONS:
Dietary Supplement: Ground beef — Ground beef naturally low in monounsaturated fatty acids or naturally high in monounsaturated fatty acids

SUMMARY:
This study tested the hypothesis that ground beef high in monounsaturated fat (MUFA) and low in saturated fat (SFA) would increase the high-density lipoprotein-cholesterol concentration and low-density lipoprotein particle diameter. In a crossover dietary intervention, 27 free-living normocholesterolemic men completed treatments in which five 114-g ground beef patties/week were consumed for 5 weeks with an intervening 4-week washout period. Patties contained 24% total fat with a MUFA:SFA ratio of either 0.71 (low MUFA, from pasture-fed cattle) or 1.10 (high MUFA, from grain-fed cattle).

DETAILED DESCRIPTION:
Participants and study design Healthy, nonsmoking males between the ages of 23 and 60 years were screened for eligibility. The 30 participants selected were not consuming restrictive diets or medications. Family histories were obtained as part of a complete physical examination that included a treadmill exercise test with an electrocardiogram. Baseline blood chemistries were analyzed by a local laboratory and all blood chemistries were within normal ranges as defined by the testing laboratory. All participants were free living and were instructed to maintain routine activities and body weight (62.2 kg of entry weight). Exercise and physical activities were not restricted, but participants were requested not to change their habitual level of physical activity. Twenty-seven of the initial 30 participants completed the study.

Of the 3 non-completers, 1 had a re-occurrence of a previous illness, another relocated, and data from the 3rd was omitted following baseline samples that showed high triglyceride concentrations (.5 mmol/L). A 2-period, randomized cross-over design was used. Each participant completed two 5-wk diet interventions in a randomly assigned order with a 4-wk washout period between the test diet interventions. The men consumed 5 ground beef patties per week for 5 wk during each dietary intervention (25 patties of each type for each ground beef intervention). The 2 interventions were low-monounsaturated fat ground beef and high-monounsaturated fat ground beef. To facilitate product distribution and blood sampling, participants were assigned to 1 of 2 groups, which were balanced with regard to age, body weight, and total cholesterol concentration at the initial screening. Group 1 began the study 2 wk before group 2. Both groups rotated through both test diets, but the pattern in which they crossed over differed between groups. Therefore, crossovers included all possible rotation sequences. Body weights were recorded weekly.

Collection and analysis of blood samples Prior to the initiation of the dietary treatments and at the end of each diet phase and after 5 minutes of seated rest, blood was collected from the participants into vacutainers from a vein in the antecubital fossa using standard phlebotomy procedures. Plasma was harvested from the blood collected with EDTA and lipoproteins preserved in plasma prior to lipoprotein separation using density gradient ultracentrifugation employing human density intervals. Determination of LDL lipoprotein diameters was by non-denaturing gradient gel electrophoresis. Particle diameters were determined by comparison with migration distances of standard proteins of known hydrated diameter. Plasma total lipoproteins isolated as the d < 1.2 kg/L fraction of plasma were separated on the basis of diameter with a gel-filtration chromatographic system to determine the relative distribution of plasma total cholesterol among very low-density lipoproteins (VLDL), LDL, and HDL lipoprotein classes. Concentrations of total cholesterol, triglycerides, and glucose in plasma were determined by separate enzymatic assays. Concentrations of serum insulin and serum C-reactive protein (CRP) were assayed using commercially available ELISA kits according to the manufacturers' instructions.

Statistical analysis We compared nutrient and dietary exchange data and final plasma glucose, lipids, insulin, CRP, and lipoprotein particle diameters to their corresponding baseline values by paired t test. Data were tested for unequal variance by the Breusch- Pagan/Cook-Weisberg test for heteroscedasticity to test the null hypothesis that the error variances were all equal. Values for changes from baseline for the low- and high-MUFA treatment groups were compared by 1-way analysis of variance, with ground beef type as the treatment effect. Associations among plasma analytes were assessed using Pearson correlation coefficients. P-values were considered significant at P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking

Exclusion Criteria:

* Consuming restrictive diets, cholesterol-lowering medications

Ages: 23 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Males
Enrollment: 27 (Actual)
Dates: Start 2006-03-27 (Actual); Primary Completion 2006-05-31 (Actual); Study Completion 2006-05-31 (Actual)

PRIMARY OUTCOMES:
Lipoprotein cholesterol | 5 weeks
  Plasma very low-density, low-density, and high-density cholesterol concentrations
Low-density lipoprotein particle size | 5 weeks
  Plasma low-density lipoprotein particle size

SECONDARY OUTCOMES:
C-reactive protein | 5 weeks
  Plasma C-reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Smith, Ph.D., Principal Investigator — Texas A&M University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gilmore LA, Walzem RL, Crouse SF, Smith DR, Adams TH, Vaidyanathan V, Cao X, Smith SB. Consumption of high-oleic acid ground beef increases HDL-cholesterol concentration but both high- and low-oleic acid ground beef decrease HDL particle diameter in normocholesterolemic men. J Nutr. 2011 Jun;141(6):1188-94. doi: 10.3945/jn.110.136085. Epub 2011 Apr 27. PMID 21525253